CLINICAL TRIAL: NCT07317622
Title: Identification and Classification of the Bereaved Population Attending Nursing Consultations in Primary Care; Proposal and Effectiveness of a Brief Intervention
Brief Title: Effectiveness of a Brief Intervention for Bereaved Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Servicio Canario de Salud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUC_2024_91
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Bereavement
Keywords: bereavement; primary care nursing; community health nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant group (Experimental)
  Interventions: Other: Facilitating Grief

INTERVENTIONS:
Other: Facilitating Grief — This intervention, called "Facilitating Grief," begins with an initial nursing assessment using the Psychosocial Nursing Diagnosis Questionnaire (PSDQ), the Relationship Continuity Scale, and an exploration of manifestations related to the grief situation. This initial assessment lasted between one and three hours, depending on the individual. Subsequently, a personalized care plan was established using standardized language, applying the most appropriate interventions for each person experiencing grief. The intervention also includes follow-up through several subsequent consultations (between two and four), in which the care plan is reviewed and adjusted according to the individual's progress, and a final assessment to evaluate the results achieved.

SUMMARY:
Grief is the response to the death of a loved one. The loss of a loved one requires a grieving process that allows one to adapt to the new situation. The main objective of this study is to identify people in a situation of bereavement who attend nursing consultations in Primary Care on the island of Tenerife, through opportunistic recruitment with the aim of carrying out a brief nursing intervention on those who are classified as being in a situation of bereavement.

DETAILED DESCRIPTION:
Grief is a complex and multidimensional process involving an emotional, cognitive, behavioral, and spiritual response to loss. From a nursing perspective, it is recognized as important to address this phenomenon holistically, considering the personal, familial, and sociocultural factors that influence its experience. According to the NANDA-I taxonomy, the diagnoses of maladaptive grief, risk for maladaptive grief, and readiness for enhanced grief fall under the coping/stress tolerance domain, reflecting the need for interventions focused on adaptation and emotional well-being.

In the healthcare setting, the primary care nurse plays a key role as the professional who maintains continuous contact with individuals and their families. The nursing intervention Facilitating Grief (NIC 5290) integrates activities such as active listening, therapeutic communication, reality orientation, music therapy, and the use of personal journals. These strategies promote emotional expression, life reorganization, and personal resilience. The use of standardized instruments (such as the Psychosocial Nursing Diagnoses Questionnaire) allows for the identification of risk factors and the planning of evidence-based care.

The proposed secondary objectives are the following: To detect risk factors that may predispose patients attending nursing consultations to maladaptive grief; To understand the usual management of people in a state of grief and their care needs; To design a brief nursing intervention in Primary Care nursing consultations and evaluate its effectiveness; and To raise awareness among Primary Care professionals about grief, its characteristics and approach, through training activities.

The null hypothesis (H0) of this research establishes that, in the studied population, brief nursing intervention does not produce a significant effect on the effectiveness of nursing care in accompanying grief or in preventing its complications.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old.
* That they answer affirmatively to at least one of the following two questions:

Have you lost a loved one in the last year? Are you grieving the loss of a loved one?

- After being informed, agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* People with language barriers.
* People with cognitive impairment.
* People with severe sensory deficits.
* People with a history of anxiety disorders, diagnosed severe depression, or other problems (emotional, coping, etc.) that prevent them from participating in the collection of information necessary for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with Clinical manifestations of their grief situation | Pre and post intervention (at 4 or 6 weeks)
  According to the defining characteristics and risk factors of NANDA-I grief diagnoses
Number of participants with Continuity of Bonds internalized or externalized | Pre and post intervention (at 4 or 6 weeks)
  The Continuity of Bonds Scale is an instrument that explores how the bereaved person continues to relate symbolically and emotionally to the deceased. It consists of 16 questions with two dimensions (internalized, 10 items, and externalized, 6 items). Responses are on a Likert scale from 1 to 4 points (1 = "not at all", 4 = "constantly").
Number of participants with Pssychosocial problems | Pre and post intervention (at 4 or 6 weeks)
  The Psychosocial Nursing Diagnosis Questionnaire (PSDN) is a validated tool. This instrument includes up to 28 psychosocial nursing diagnoses, grouped into six dimensions: health perception/management, behavior/social interaction, emotional/self-perception, caregiver burden, loss/grief, and body image disturbance. It uses Likert-type scales and dichotomous questions to grade responses, assigning different diagnostic labels based on predefined combinations.
Number of participants willing to improve their grief | Pre and post intervention (at 4 or 6 weeks)
  Nursing diagnosis " Readiness for enhanced grief " (Yes/No) and presence/absence of the following defining characteristics: Desire to carry on the deceased's legacy; Desire to engage in previous activities; Desire to enhance grief coping; Desire to enhance forgiveness; Desire to enhance hope; Desire to enhance personal growth; Desire to enhance sleep-wake cycle; Desire to integrate feelings of anger; Desire to integrate feelings of despair; Desire to integrate feelings of guilt; Desire to integrate feelings of remorse; Desire to integrate positive feelings; Desire to integrate positive memories of the deceased; Desire to integrate the possibilities of a happy life; Desire to integrate the possibilities of a meaningful life; Desire to integrate the possibilities of a purposeful life; Desire to integrate the possibilities of a satisfying life; Desire to integrate the loss; Desire to invest energy in new interpersonal relationships.
Number of participants with maladaptive grief | Pre and post intervention (at 4 or 6 weeks)
  Nursing diagnosis " maladaptive grief " (Yes/No) and presence/absence of the following defining characteristics: Anger; Anxiety Decreased performance in life roles; Depressive symptoms; Distress over the deceased; Excessive stress; Feelings of emptiness; Avoidance of grief Non-acceptance of death; Persistent painful memories; Preoccupation with thoughts about the deceased person; Rumination (obsessive ideas) about the deceased person; Searching for the deceased person; Self-blame.
Number of participants at risk of maladaptive grief | Pre and post intervention (at 4 or 6 weeks)
  Nursing diagnosis " risk of maladaptive grief " (Yes/No) and presence/absence of the following defining characteristics: Difficulty dealing with recurrent crises; Excessive emotional disturbance; Inadequate social support; Anxious attachment (in their relationship with others); Avoidant attachment (in their relationship with others).

SECONDARY OUTCOMES:
Number of participants with chronic health problems | Pre-intervention
  Dichotomous variables (Yes/No)
Number of participants receiving pharmacological treatment | Pre-intervention
  Dichotomous variables (Yes/No)
Number of caregiver participants | Pre-intervention
  Dichotomous variables (Yes/No)
Time since death | Pre-intervention
  Continuous quantitative variable (days, months, years)
Cause of death | Pre-intervention
  Nominal qualitative variable

CONTACTS AND LOCATIONS:
Locations (1):
- Gerencia Atención Primaria Tenerife, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Undecided